CLINICAL TRIAL: NCT03896438
Title: Increased Thalamocortical Connectivity in Tdcs-potentiated Generalization of Cognitive Training
Brief Title: Maximizing the Impact of Neuroplasticity Using Transcranial Electrical Stimulation Study 2
Acronym: MINUTES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCH-2018-26586_02; 1RF1MH116987-01 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Transcranial Direct Current Stimulation; Schizophrenia; Schizoaffective Disorder
Keywords: tDCS; cognitive training; functional connectivity
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- right active-tDCS (Experimental): 2-3 times/week for 12 weeks: ramp-up for 30 seconds, 2mA right (AF4 anode - AF3 cathode) for 20 min, and then ramp-down for 30 seconds.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- left active-tDCS (Experimental): 2-3 times/week for 12 weeks: ramp-up for 30 seconds, 2mA left (AF3 anode - AF4 cathode) for 20 min, and then ramp-down for 30 seconds.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- sham tDCS (Sham Comparator): Current will be turned off immediately after the initial 30-second ramp-up period.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Three different stimulation montages will be programmed: right, left and sham. During the Ramp periods, 2 mA current will be delivered to both AF3 and AF4 with an ascending (RampUp) and descending ramp (RampDown) over 30 sec via two saline soaked electrode sponges (~ 25cm²; current density = 0.08 mA/cm²). In this way, all subjects experience the same sensation on both sides to blind them to condition. During the Constant period, current will be set based on the Condition: Right - 2mA AF4 anode-AF3 cathode; Left - 2mA applied to AF3 anode-AF4 cathode; Sham - current turned off.

SUMMARY:
Non-invasive neuromodulation, such as transcranial direct current stimulation ( tDCS) , is emerging as an important therapeutic tool with documented effects on brain circuitry, yet little is understood about h ow it changes cognition. In particular, tDCS may have a critical role to play in generalization, that is how training in one domain generalizes to unlearned or unpracticed domains. This problem has resonance for disorders with cognitive deficits, such as schizophrenia.

Understanding how tDCS affects brain circuity is critical to the design and application of effective interventions, especially if the effects are different for healthy vs. psychiatric populations. In previous research, one clue to the mechanism underlying increased learning and generalization with tDCS was provided by neuroimaging data from subjects with schizophrenia undergoing cognitive training where increases in thalamocortical (prefrontal) functional connectivity (FC) predicted greater generalization.

The premise of this proposal is that increases in thalamocortical FC are associated with the generalization of cognitive training, and tDCS facilitates these increases. The overarching goals of this proposal are to deploy neuroimaging and cognitive testing to understand how tDCS with cognitive training affect thalamocortical circuitry in individuals with and without psychosis and to examine variability in response within both groups.

Study 1(NCT03896425) will compare right prefrontal, left prefrontal and sham tDCS during concurrent cognitive training over 12 weeks in 90 healthy controls. Study 2 will be similar in all aspects but will examine 90 patients with schizophrenia or schizoaffective disorder and include clinical assessments. Results of the study will provide crucial information about location of stimulation, length of treatment, modeled dosage, trajectory and durability needed to guide future research and interventions for cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide consent and comply with study procedures.
2. Age 18 - 60 years old.
3. Estimated IQ range within the range: 70 ≤ IQ ≤ 115.
4. Schizophrenia or schizoaffective disorder as assessed by the MINI (Mini International Neuropsychiatric Interview)(Sheehan et al., 1998).
5. Not having a current addictive disorder as measured by MINI (Mini International Neuropsychiatric Interview), or a sleep disorder.
6. Ability to participate in three weekly 45' training sessions over 12 weeks and participate in four assessments.
7. Clinically stable and on stable medications for at least one month before start of study.

Exclusion Criteria:

1. Any medical condition or treatment with neurological sequelae (e.g. stroke, tumor, loss of consciousness > 30 min, HIV).
2. Contraindications for tDCS or MRI scanning (tDCS contraindication: history of seizures; MRI contraindications: The research team will utilize the CMRR Center's screening tools and adhere to the screening SOP during enrollment of all research participants in this protocol. The CMRR Center's screening tools and SOP are IRB approved under the CMRR Center Grant (HSC# 1406M51205) and information regarding screening procedures is publicly available on the CMRR website (CMRR Policies / Procedures).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants dropped out before randomization, but completed the baseline session. Due to difficulty with recruitment and retention that led to low numbers, we were unable to conduct any statistical analyses. In addition, two participants were removed from the DPX neuroimaging results due to motion artefacts. One participant was removed from the NBack neuroimaging results due to scanning issues. One participant was removed from UPSA analyses due to missing scores.
Period: Overall Study
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
Started | 1 | 4 | 4
Completed | 0 | 1 | 2
Not Completed | 1 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS | Total
Number analyzed (Participants) | 1 | 4 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (0) | 33 (14.28) | 42 (6.48) | 36.11 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 5
  Male | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 2 | 3 | 6
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Changes in Thalamocortical Functional Connectivity (FC)
Description: Most participants completed MRI sessions on a 3T scanner located in the Center for Magnetic Resonance Research (CMRR) at the University of Minnesota. FC measures how different brain regions change in activation together. We characterized FC using global connectivity from graph theory analysis. We extracted the fMRI time courses from 454 parcellations defined by the 400 S4 Schaefer Atlas (Schaefer et al., 2018) combined with the Melbourne Subcortex Atlas (Tian et al., 2020). We computed the absolute value of the Pearson's correlation for all possible pairs of time series, creating a 454x454 (N x N) connectivity matrix, which was then reduced to 10% most significant connections by subject. We estimated the FC by calculating the node strength for each parcellation, which is the weighted mean of all significant connections, from these connectivity matrices. Finally, we averaged node strength across parcellations to calculate global node strength. Higher values indicate more brain-wide FC.
Time Frame: baseline
Population: We had difficulty with recruitment, so there were zero people that completed the right active-tDCS for this attribute, and therefore we cannot report anything for the mean (there is no value)
Measure: Mean (Standard Deviation); unit: a.u.
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 3 | 0
a.u. | 18.2 (3) | 17.3 (1.7) |

2. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the N-back Task.
Description: Task-dependent thalamocortical connectivity associated with the N-back task was calculated by modeling the block task design together with the thalamic regressor using psychophysiological interaction analysis (PPI). The thalamic regressor is the time series of the mediodorsal thalamus from the Melbourne atlas. The primary analysis focused on the 2-back conditions alone. The PPI analysis calculates the functional connectivity between the mediodorsal thalamus and all other brain regions specifically during 2-back trials. Neural activation related to the thalamic regressor was compared to neural activation during the fixation (no choices made) to normalize the relative activation (z-score). Positive values indicate increased functional connectivity with the thalamus during the 2-back choices. A z-score of zero represents no difference compared to the fixation cross (no choices). We report the average z-score of the PPI regressor within the control network (Yeo et al., 2011).
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 0
z-score | 0.02 (0.39) | -0.21 (0.27) |

3. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the DPX Task.
Description: Task-dependent thalamocortical connectivity associated with the Dot Pattern Expectancy (DPX) task demands will be identified by analyzing cue and probe events together with the thalamic regressor using psychophysiological interaction analysis (PPI). The thalamic regressor is the time series of the mediodorsal thalamus from the Melbourne atlas. We examined B-cue related connectivity. The PPI analysis calculates the functional connectivity between the mediodorsal thalamus and all other brain regions specifically during B-cue trials. Neural activation related to the thalamic regressor was compared to neural activation during the fixation (no choices made) to normalize the relative activation (z-score). Positive values indicate increased functional connectivity with the thalamus during the B-cue responses. A z-score of zero represents no difference compared to the fixation cross (no choices). We report the average z-score of the PPI regressor within the control network.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 1
z-score | -0.02 (0.37) | -0.03 (0.58) | 0.45 (0)

4. Primary Outcome: Change in N-back Performance
Description: The n-back task measures working memory capacity. The participant is presented with a series of stimuli and instructed to indicate with a button press when the current stimulus matches the stimulus that appeared a pre-determined number (n) of trials before. d' (d prime) will be calculated as a measure of signal detection, which indicates the normalized rate of hits to false positives (d' = z(H) - z(F)). Increase in d' signifies improved signal detection, i.e. a better outcome. A d' near zero indicates a performance at chance, i.e., a poor performance. The range is -4.65 to 4.65
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: d-prime score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 1
d-prime score | 1.99 (0.95) | 1.45 (0.31) | 0 (0)

5. Primary Outcome: Change in DPX Performance
Description: The Dot Pattern Expectancy (DPX) task is an adaptation of the expectancy AX task that uses pairs of simple dot patterns rather than letter pairs as stimuli. The DPX task will be performed in 3 blocks. Each trial consists of a cue dot pattern followed by a probe dot pattern. Different combinations of cues and probes enable the identification of a specific deficit in a subject's ability to maintain goal-relevant information throughout a trial. Timing will be jittered and each block of the DPX task will consist of 40 trials: 24 AX (60%), 6 AY (15%), 6 BX (15%) and 4 BY (10%). Each block will last 6 minutes. d'-context will be calculated as a measure of signal detection, which indicates the normalized rate of AX hits to BX false positives (d' = z(H) - z(F)). Increase in d' -context signified improved signal detection, i.e. a better outcome. A d' near zero indicates a performance at chance, i.e., a poor performance. The range is -4.65 to 4.65.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: d-prime score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 1
d-prime score | 2.78 (0.73) | 2.65 (0.72) | 2.51 (0)

6. Primary Outcome: Change in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: Intends to provide a relatively brief evaluation of key cognitive domains relevant to schizophrenia and related disorders. The composite score is reported as a T-score, with a mean of 50 and standard deviation of 10. Higher values indicate greater cognitive functioning.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Right Active tDCS: 2-3 times/week for 12 weeks: ramp-up for 30 seconds, 2mA right (AF4 anode - AF3 cathode) for 20 min, and then ramp-down for 30 seconds.
  Transcranial Direct Current Stimulation (tDCS): Three different stimulation montages will be programmed: right, left and sham. During the Ramp periods, 2 mA current will be delivered to both AF3 and AF4 with an ascending (RampUp) and descending ramp (RampDown) over 30 sec via two saline soaked electrode sponges (~ 25cm²; current density = 0.08 mA/cm²). In this way, all subjects experience the same sensation on both sides to blind them to condition. During the Constant period, current will be set based on the Condition: Right - 2mA AF4 anode-AF3 cathode; Left - 2mA applied to AF3 anode-AF4 cathode; Sham - current turned off.
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active tDCS
Number analyzed (Participants) | 4 | 4 | 1
T-score | 53 (9.7) | 48.8 (11.9) | 48 (0)

7. Primary Outcome: Changes in Thalamocortical Functional Connectivity (FC)
Description: as for outcome 1
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 3 | 0
arbitrary units | 18.8 (2.7) | 17.4 (2.4) |

8. Primary Outcome: Changes in Thalamocortical Functional Connectivity (FC)
Description: as for outcome 1
Time Frame: post-test (week 12)
Population: We had difficulty with recruitment, so there were zero people that completed the right and left active-tDCS for this attribute, and therefore we cannot report anything for the mean (there is no value)
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 0 | 2 | 0
arbitrary units |  | 16.5 (3.2) |

9. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the N-back Task.
Description: as for outcome 2
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 2 | 0
z-score | -0.03 (0.58) | -0.92 (0.63) |

10. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the N-back Task.
Description: as for outcome 2
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 2 | 1 | 0
z-score | -0.38 (0.01) | -1.24 (0) |

11. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the DPX Task.
Description: PPI regressor (z-score) within Control Network associated with B-cue Task-dependent thalamocortical connectivity associated with the DPX task demands will be identified by analyzing cue and probe events together with the thalamic regressor using psychophysiological interaction analysis (PPI). The thalamic regressor is the time series of the mediodorsal thalmus from the Melbourne atlas (THA-DAm; Tian et al., 2020). Preliminary analysis for the DPX task will examine B-cue related connectivity alone. We report the average z-score of the PPI regressor within the control network (Yeo et al., 2011). Neural activation was normed to calculated z-scores, such that postive values indicate increased connectivity with the thalamus, and negative values indicate decreased connectivity with the thalamus.
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 1 | 0
z-score | -0.14 (0.16) | -0.52 (0) |

12. Primary Outcome: Changes in Task-dependent Thalamocortical Functional Connectivity (fMRI) During the DPX Task.
Description: as for outcome 11
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 2 | 1 | 0
z-score | 0.04 (0.23) | 0.47 (0) |

13. Primary Outcome: Change in N-back Performance
Description: as for outcome 4
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: d-prime score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 3 | 0
d-prime score | 2.71 (1.13) | 2.31 (0.61) |

14. Primary Outcome: Change in N-back Performance
Description: as for outcome 4
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: d-prime score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 2 | 1 | 0
d-prime score | 3.81 (0.58) | 1.81 (0) |

15. Primary Outcome: Change in DPX Performance
Description: as for outcome 5
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: d-prime score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 2 | 0
d-prime score | 3.42 (0.44) | 3.48 (0.08) |

16. Primary Outcome: Change in DPX Performance
Description: as for outcome 5
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: d-prime score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 2 | 1 | 0
d-prime score | 3.68 (0.11) | 1.57 (0) |

17. Primary Outcome: Change in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: MCCB Composite T-Score Intends to provide a relatively brief evaluation of key cognitive domains relevant to schizophrenia and related disorders. The composite score is reported as a T-score, with a mean of 50 and standard deviation of 10. Higher values indicate greater cognitive functioning.
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active tDCS
Number analyzed (Participants) | 3 | 3 | 0
T-score | 48.33 (8.5) | 49.7 (18.6) |

18. Primary Outcome: Change in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 17
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active tDCS
Number analyzed (Participants) | 1 | 2 | 0
T-score | 42 (0) | 69.5 (4.9) |

19. Primary Outcome: Change in Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) Composite Score
Description: as for outcome 17
Time Frame: follow-up (week 24)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active tDCS
Number analyzed (Participants) | 0 | 2 | 0
T-score |  | 68 (2.8) |

20. Secondary Outcome: Change in University of California San Diego Performance-Based Skills Assessment - Brief (UPSA-B)
Description: Measures functional capacity by assessing skills involved in everyday tasks important to daily living. Points are scored for each of two sub scales based on the participant's correct performance of items in the sub scale (incorrect: 0 points, correct: 1 or 2 points). Points are used to derive a sub scale score by dividing points scored by the number of items in the sub scale (percentage correct) and multiplied by 50. The two sub scale scores are then added to derive the total score, with a possible range of 0-100. Higher scores represent better outcomes.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 3 | 1
raw score | 85.5 (7.9) | 76.3 (6.8) | 84 (0)

21. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Score
Description: Measures symptom severity in patients with schizophrenia. Scores are assigned for symptom categories based on a semi-structured clinical interview with anchored severity scales (1-7) for each symptom category. Total score is derived by adding up individual symptom scores, resulting in a total score range of 24-168. Higher scores indicate greater symptom severity. A decrease in scores over time would indicate symptom reduction, i.e. a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 1
raw score | 51.5 (9.7) | 53.3 (8.5) | 33 (0)

22. Secondary Outcome: Change in Brief Negative Symptom Scale (BNSS) Score
Description: Measures of symptom severity in patients with schizophrenia with an emphasis on negative symptoms. Scores are assigned to symptom categories based on a semi-structured clinical interview with anchored severity scales (0-6 or 0-9). Total score is derived by adding up individual symptom scores, resulting in a total score range of 0-90. Higher scores indicate greater symptom severity. A decrease in scores over time would indicate symptom reduction, i.e. a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 1
raw score | 9.25 (7.04) | 12.5 (10.7) | 5 (0)

23. Secondary Outcome: Change in University of California San Diego Performance-Based Skills Assessment - Brief (UPSA-B)
Description: as for outcome 20
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 3 | 0
raw score | 83 (4.3) | 61.3 (7.1) |

24. Secondary Outcome: Change in University of California San Diego Performance-Based Skills Assessment - Brief (UPSA-B)
Description: as for outcome 20
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 1 | 2 | 0
raw score | 80 (0) | 82.5 (3.5) |

25. Secondary Outcome: Change in University of California San Diego Performance-Based Skills Assessment - Brief (UPSA-B)
Description: as for outcome 20
Time Frame: follow-up (week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 1 | 2 | 0
raw score | 85 (0) | 74.5 (7.8) |

26. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Score
Description: as for outcome 21
Time Frame: mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 3 | 0
raw score | 55 (9) | 49 (8.2) |

27. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Score
Description: as for outcome 21
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 1 | 2 | 0
raw score | 50 (0) | 40.5 (4.9) |

28. Secondary Outcome: Change in Brief Psychiatric Rating Scale (BPRS) Score
Description: as for outcome 21
Time Frame: follow-up (week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 1 | 2 | 0
raw score | 37 (0) | 30 (5.6) |

29. Secondary Outcome: Change in Brief Negative Symptom Scale (BNSS) Score
Description: as for outcome 22
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 4 | 4 | 1
raw score | 9.25 (7.04) | 12.5 (10.7) | 5 (0)

30. Secondary Outcome: Change in Brief Negative Symptom Scale (BNSS) Score
Description: as for outcome 22
Time Frame: Mid-test (week 6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 3 | 3 | 0
raw score | 7.3 (6.8) | 14 (8.9) |

31. Secondary Outcome: Change in Brief Negative Symptom Scale (BNSS) Score
Description: as for outcome 22
Time Frame: post-test (week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 1 | 2 | 0
raw score | 20 (0) | 12.5 (10.6) |

32. Secondary Outcome: Change in Brief Negative Symptom Scale (BNSS) Score
Description: as for outcome 22
Time Frame: follow-up (week 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Left Active-tDCS | Sham tDCS | Right Active-tDCS
Number analyzed (Participants) | 1 | 2 | 0
raw score | 13 (0) | 17 (11.3) |

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Right Active-tDCS | Left Active-tDCS | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 3/4 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Right Active-tDCS (N=1) | Left Active-tDCS (N=4) | Sham tDCS (N=4)
Burn from tDCS electrode (General disorders) | 0 (0) | 1 (1) | 0 (0)
Reported brain fog(moderate or greater) (General disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03896438/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03896438/ICF_001.pdf